CLINICAL TRIAL: NCT05718219
Title: A Phase I, First-in-Human, Open-Label Study to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0348 in Subjects With Advanced Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0348 in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0348-101
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1A ( SIM0348 Monotherapy) (Experimental): Part 1A (dose escalation and dose expansion) Cohorts of at least 3 participants each will be treated with escalating doses of SIM0348 alone or in combination with Sintilimab . Dose expansion part will be decided based on the findings of dose escalation part. Part 1A was to evaluate single agent SIM0348 once weekly or once every 3 weeks.
  Interventions: Drug: SIM0348
- Part 1B (SIM0348 + Sintilimab ) (Experimental): Part 1B (dose escalation and dose expansion) Cohorts of at least 3 participants each will be treated with escalating doses of SIM0348 alone or in combination with Sintilimab. Dose expansion part will be decided based on the findings of dose escalation part. In Part 1B, selected dose from Part 1A were evaluated in Part 1B when they were combined with Sintilimab (200mg once every 3 weeks)
  Interventions: Drug: SIM0348 + Sintilimab
- Part 2A (SIM0348 Monotherapy Cohort Expansion) (Experimental): Selected doses from Part 1A will be evaluated for SIM0348 administered as a single agent. SIM0348 will be given via IV infusion until disease progression or loss of clinical benefit.
  Interventions: Drug: SIM0348
- Part 2B (SIM0348 + Sintilimab Cohort Expansion) (Experimental): Selected doses from Part 1B will be evaluated for SIM0348 when they were combined with Sintilimab (200mg once every 3 weeks)
  Interventions: Drug: SIM0348 + Sintilimab

INTERVENTIONS:
Drug: SIM0348 — Several dose levels will be evaluated for SIM0348 administered as a single agent . SIM0348 will be given via IV infusion on Day 1, Day 8, Day 15, Day 22 of each cycle (28-day or depending on study cohort and phase) until disease progression or loss of clinical benefit.
  Arms: Part 1A ( SIM0348 Monotherapy); Part 2A (SIM0348 Monotherapy Cohort Expansion)
Drug: SIM0348 + Sintilimab — Selected doses from Part 1A will be evaluated for SIM0348 when they were combined with Sintilimab (200mg once every 3 weeks).
  Arms: Part 1B (SIM0348 + Sintilimab ); Part 2B (SIM0348 + Sintilimab Cohort Expansion)

SUMMARY:
This is a multicenter, open label, phase I trial to evaluate the safety and tolerability, pharmacokinetic/ pharmacodynamic characteristics and to assess the preliminary efficacy of SIM0348 as monotherapy or with sintilimab in adult subjects with advanced and metastatic solid tumors. The trial starts with a dose escalation and dose expansion part (Part 1) followed by a cohort expansion part (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Must have failed at least one established standard anti-cancer therapies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy at least 12 weeks
* Adequate hematologic and end organ function
* Histologic documentation of locally advanced, recurrent, or metastatic incurable malignancy that has progressed after at least one available standard therapy; or for which standard therapy has proven ineffective, intolerable, or considered inappropriate; or for which a clinical trial of an investigational agent is a recognized standard of care
* Confirmed availability of representative tumor specimens
* Measurable disease according to RECIST Version 1.1

Exclusion Criteria:

* Malignancies other than disease under study within 2 years prior to Day 1 of Cycle 1
* Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases
* History of interstitial lung disease, evidence of active pneumonitis (history of radiation pneumonitis in the radiation field [fibrosis] is permitted), and active pneumonia that are considered inappropriate by the investigator
* History of severe hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of autoimmune disease
* Positive human immunodeficiency virus (HIV) test
* Severe infection within 2 weeks prior to the first dose of study treatment
* Significant cardiovascular disease
* History of allogeneic tissue/solid organ transplant or graft-versus-host disease
* Known clinically significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Dose-limiting toxicity (DLT) | DLT evaluation window was from Baseline to the end of Cycle 1 (up to 28 days)
Part 2: Objective response rate (ORR) assessed by Investigator per RECIST v.1.1 | up to approximately 2 years
  To evaluate the anti-tumor activity of SIM0348 alone and in combination with Sintilimab

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No